CLINICAL TRIAL: NCT02857829
Title: The Effects of a Combination of Nootropic Ingredients on Cognition in Healthy Young Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nootrobox, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Nootrobox_Maastricht
Record Dates: First submitted 2016-07-30; First posted 2016-08-05 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Biomedical Enhancement
Keywords: Cognition; working memory; nootropic; reaction time; healthy individuals; cognitive enhancement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Caffeine-alone (Active Comparator): The effects of the combination will be compared to both placebo and caffeine-alone, to test the hypothesis that the blend of ingredients will enhance cognitive measures greater than the most commonly used cognitive enhancer, caffeine.
  Interventions: Dietary Supplement: Caffeine-alone
- CAF+ (Experimental)
  Interventions: Dietary Supplement: CAF+

INTERVENTIONS:
Dietary Supplement: CAF+ — CAF+ will be a blend consisting of caffeine (100 mg), L-theanine (200 mg), vinpocetine (40 mg), L-tyrosine (300 mg), pyridoxine (1 mg), and cobalamin (20 mg).
  Arms: CAF+
Dietary Supplement: Caffeine-alone — Caffeine (100 mg)
  Arms: Caffeine-alone
Other: Placebo — Rice flour
  Arms: Placebo

SUMMARY:
Achieving optimal concentration during cognitively demanding tasks is of immense human value. Despite our understanding of the important role that attention, working memory, and fluid intelligence play in professional success, and the huge individual differences in these constructs, the modulation of these cognitive domains has not been rigorously studied. From the widespread use of caffeine, to the more questionable and increasing use of prescription medications to achieve peak attention, the tremendous interest in achieving cognitive performance has driven individuals to experiment, often with prescription and illegal drugs. Herein, we aim to standardize and extend the study of attention modulating substances, to identify blends that achieve safe enhancements in attention and working memory. Specific to this proposal, we aim to develop CAF+, a blend of natural and generally regarded as safe compounds to improve attention and working memory in normal, healthy individuals. CAF+ is composed of caffeine (100 mg), L-theanine (200 mg), vinpocetine (40 mg), L-tyrosine (300 mg), pyridoxine (0.06 mg), and cobalamin (20 mg).

DETAILED DESCRIPTION:
Rationale: There is still a great need to find treatments that can improve cognitive function in people that suffer from memory and attention problems, as well as healthy, young individuals. There are various natural ingredients that have been claimed to improve cognitive functions in humans (e.g., caffeine, L-theanine, vinpocetine). These ingredients have a different mechanism of action and are assumed to have a general effect on brain function. It is hypothesized that a combination of these natural ingredients may be more effective to improve cognitive performance. In this study we would like to test the cognition-enhancing potential of a mixture of different natural ingredients.

Objective: Examine the effects of a treatment that consists of different natural ingredients on cognitive performance in young healthy subjects. These effects will be compared with caffeine treatment, a natural ingredient that has been found to improve cognition in various studies.

Study design: This study will use a double-blind placebo controlled, cross-over design.

Study population: Twenty-one healthy subjects in the age range from 18-35 years will be included.

Intervention: The subjects will be tested three times. At each test session they will receive one capsule (Placebo, Caffeine, or CAF+).

Main study parameters/endpoints: The primary outcome measure is the number of recalled words in a verbal word learning task.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The subjects who will be included in the study will visit the testing site four times (medical screening + practice session, and three test sessions). Each testing session will last 2.5 h. In total the subjects will spent about 10 h when they participate. During the three test sessions the subjects will receive a capsule that contains a placebo, caffeine or a combination of different natural ingredients. These treatments are well tolerated. No adverse reactions of treatment are expected. The subjects have to abstain from drinking coffee and smoking the evening before the test days. The results of this study will reveal whether a combination of different natural ingredients is more effective than coffee to improve cognitive functions. In the light of a great demand for finding treatments that can be beneficial for old subjects suffering from age-related cognitive impairments, it is considered that the risks are minimal and there is a considerable potential benefit.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-30
* Willing to sign informed consent

Exclusion Criteria:

* Suffer from or have a history of cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal, haematological or psychiatric illness (Also those volunteers who have a first-degree relative with a psychiatric disorder or a history with a psychiatric disorder will be excluded)
* Alcohol consumption >20 drinks/week
* pregnant or lactating
* use of medication of than oral contraceptives
* use of recreation drugs 2 weeks before until the end of the experiment
* any motor or sensory deficits which could reasonably be expected to affect test performance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Verbal Memory: Immediate recall score | Up to 12 weeks
  Verbal Memory will be assessed by an adjusted version of the Rey Auditory Verbal Learning Test (Lezak, 1995): the visual verbal learning test (Riedel, Klaassen, Deutz, van Someren, & van Praag, 1999). This test consists of a list of 30 Dutch monosyllabic words (18 nouns, 12 adjectives) of which subjects have to remember as many as possible. All words are presented one by one on a computer screen, in three trials with the same item sequence. After each trial, the subjects are asked to name as many words as they can (immediate recall). Thirty minutes after the third trial, the subject is requested to recall as many words as possible (delayed recall). Next to the delayed recall, a recognition test will be assessed, consisting of all former and 30 comparable new words. Subjects are asked to respond whether they have seen the word during the learning trials by means of pressing a "yes" or a "no" button.

SECONDARY OUTCOMES:
Verbal Memory: Delayed recall score | Up to 12 weeks
  Thirty minutes after the third trial of the Verbal Learning Task, the subject is requested to recall as many words as possible (delayed recall). Next to the delayed recall, a recognition test will be assessed, consisting of all former and 30 comparable new words. Subjects are asked to respond whether they have seen the word during the learning trials by means of pressing a "yes" or a "no" button.
Working memory | Up to 12 weeks
  Working memory will be assessed by the n-back task. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. The load factor n can be adjusted to make the task more or less difficult. In this study, we use a 0-back, 1-back and 2-back task, in which the 0-back is a simple focused attention/speed task and the 1- and 2-back require accessing information from working memory.
Response inhibition and focused attention | Up to 12 weeks
  The Stroop task will be used for this measure. It is well known for its ability to induce interference, and assesses response inhibition and focused attention. In this task, colour names (in Dutch) are printed in coloured ink; in the congruent category, the colour name and the colour of the ink are the same, in the incongruent category they are not. The subjects have to name the colour of the ink, not the words themselves. However, because of the urge to read the printed words (even if one is asked to ignore them) interference occurs. Since the printed words and ink colour differ in the incongruent category, interference is larger in this category than in the congruent category; this is called the 'Stroop effect' and is known to remain even after extended practices. The colours used in this task are in blue, red, green and yellow. The colour of the ink has to be named by pressing one out of four buttons, which each represent one of the colours.
Complex-scanning and visual tracking | Up to 12 weeks
  The digit-symbol substitution task will be used for this measure as follows: The screen shows a series of 9 numbered symbols that represent a "key" The participant is then presented with a series of parallel boxes that contain a symbol in the top half of the box. He or she must provide a "number" response for the bottom half by referring to the key. The score is calculated by how many corrects responses can be made within 90 s.
Simple and -choice reaction time | Up to 12 weeks
  The task is divided into two parts. First the participant must react as soon as the button enlightens in the centre of the response box, by pressing that button. In the second part one of three possible buttons will light up. The participant is instructed to respond as quickly as possible.

OTHER OUTCOMES:
Heart Rate | Up to 12 weeks
Blood Pressure | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arjan Blokland, PhD, Principal Investigator — Maastricht University; Anke Sambeth, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No